## Statistical Analysis Plan

Unique Protocol ID: STUDY20190922

## NCT05469438

Brief Title: IMAS Optimization and Applicability in Acute and Subacute Stroke.

Official Title: IMAS Optimization and Applicability in Acute and Subacute Stroke.

Document Date: January 2, 2019

## Data Analysis Plan

| We determined the sample size (recruitment up to 60 subjects for n=30 subjects completing the protocol) based on: 1. A sample size of N=15 patients provides at least 80% power (alpha=0.05) to detect a mean difference of 3% in arm movement mean speed, 2.7% in arm movement mean peak speed, and 2.5% in arm movement jerk between an affected and non-affected limb. |
|---|
| hen, we will assess |
| a broad class of generalized linear models to predict disease features and ability to recover as a function |
| of the signals acquired from the sensor suite. |
| We will then assess |
| if our computational algorithms can predict a patient's FM score and a patient's motor recovery state |

after rehabilitation.